CLINICAL TRIAL: NCT01762644
Title: A Phase IIB/III Multicenter Randomized Trial to Evaluate the Combination of Low-Dose Cyclosporine and Omeprazole Versus Omeprazole Alone in Participants With New Onset Type 1 Diabetes.
Brief Title: The Insulin Independence Trial (IIT) Evaluating the Safety and Efficacy of Oral Cyclosporine and Oral Omeprazole for Insulin Independence Among Recent Onset Type 1 Diabetes Patients
Acronym: IIT
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was withdrawn prior to enrollment.
Sponsor: Perle Bioscience, Inc. (Industry)
Collaborators: Syreon Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRL001-PB-01; 2015-000105-39 (EudraCT Number)
Record Dates: First submitted 2013-01-02; First posted 2013-01-08 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2015-07

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Insulin Independence; Beta Regeneration; Immune Tolerance Agent; Omeprazole; Cyclosporine
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Cyclosporine; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Immune Tolerance and Proton Pump Inhibitor
  Interventions: Drug: Oral Cyclosporine and Oral Omeprazole
- Arm 2 (Active Comparator): Proton Pump Inhibitor
  Interventions: Drug: Oral Omeprazole

INTERVENTIONS:
Drug: Oral Cyclosporine and Oral Omeprazole
  Arms: Arm 1
Drug: Oral Omeprazole
  Arms: Arm 2

SUMMARY:
The purpose of this study is to determine if the combination of oral cyclosporine, an immune therapy and oral omeprazole, a proton pump inhibitor, are effective in rendering insulin independence among recent onset type 1 diabetes patients. This two-arm study is designed to evaluate the safety and efficacy for insulin independence of two FDA and EMA-approved therapies among recent onset type 1 diabetes patients.

One of the greatest new insights of today in the field of type 1 diabetes, is the understanding that in man, unlike the success seen in type 1 diabetes mouse models, there is no beta cell regeneration with immune therapy alone. In man, type 1 diabetes is now considered to be a disease of both autoimmunity and lack of beta cell regeneration (Levetan 2103).

More than 500 patients with new onset type 1 diabetes have been given cyclosporine and some studies have demonstrated as high as a 57% insulin-free remission rate that was not sustained due to the lack of beta cell regeneration (Feutren 1986, Bougneres 1988, Eisenbarth 1989, Sobel 2010). Studies among diabetes patients with proton pump inhibitors have shown the potential to increase beta cell mass by 40%, but among type 1 patients without immune protection, such outcomes cannot be not achieved (Singh 2012, Griffin 2014).

The usage of a beta cell regeneration agent such as omeprazole, in combination with an immune tolerance, like cyclosporine, provides both the potential ability to maintain and regenerate beta cells. This is a new paradigm for the treatment of new onset type 1 diabetes.

More than 60 human trials have been conducted among type 1 diabetes with a variety of different therapies aimed at preventing autoimmune attack on insulin-producing beta cells. None have been as effective as cyclosporine in both slowing the decline in beta cell mass and resulting in the potential for insulin-free remissions. (Canadian-European Randomized Control Trial 1988, Eisenbarth 1989, Skyler 1992, Sobel 2010).

Because cyclosporine is known for its potential side-effects, most notably in the kidney, all previous studies among type 1 patients have carefully monitored kidney function. Follow-up studies for up to 13 years among 285 type 1 patients utilizing cyclosporine for 20 months did not demonstrate renal or other side effects at the dosages that will be used in this trial (Assan 2002).

The most effective initiating dosage for insulin independence in the cyclosporine trials was 7.5 mg/kg/day, but for safety, this study will begin at a lower dosage of 5 mg/kg/day and will monitor kidney function and cyclosporine levels initially on a weekly basis. This study will use only those dosages of cyclosporine that have not demonstrated toxicity to the kidney or resulted in non-reversible side effects among more than 500 patients with recent onset type 1 diabetes treated with cyclosporine.

Omeprazole has been shown to significantly increase gastrin levels which is associated with increased beta cells. Lansoprazole has also been shown to be safe among patients with new onset type 1 diabetes for one year with a trend toward increased beta cell mass among patients with higher gastrin levels.

In a randomized trial for 12 weeks among 56 patients undergoing pancreatectomy, those randomized to receive a proton pump inhibitor had significantly increased gastrin levels, higher insulin levels and improved endocrine function by glucose tolerance testing and less pancreatic atrophy as measured by CT scans (Jang 2003).

The recently completed REPAIR T1D trial among newly diagnosed type 1 patients used a proton pump inhibitor and GLP-1 therapies for 1 year for beta regeneration failed to meet its endpoint of increased stimulated C-peptide. Lack of maintenance or regeneration of beta cells was specifically noted to have likely been due to lack of usage of immune therapy to protect beta cells (Griffin 2014, Rigby 2014).

Those patients in REPAIR T1D, who did achieve gastrin and GLP-1 levels above those in the control group had a trend towards improved preservation of C-peptide with a suggestion of a decreased rate of fall of C-peptide through 12 months (Griffin 2014 Appendix Supplemental data). Glucose levels also trended lower than controls in the intervention arm with gastrin levels above the control arm (Griffin 2014 Appendix Supplemental data). In humans, the newly forming beta cells are under the greatest immune attack among type 1 patients (Meier 2006). REPAIR T1D underscores the importance for both immune therapy with a regeneration therapy among type 1 patients (Griffin 2014, Rigby 2014).

The combination of cyclosporine with a proton pump inhibitor has the potential to demonstrate maintenance and expansion of residual beta cells. This combination therapy provides the unique ability for patients to become insulin independent.

For a request of references, please email info@perlebioscience.com

ELIGIBILITY:
Inclusion Criteria

Participants included in this study are those who meet all of the following criteria:

1. Male or female participant 10-20 years old.
2. Diagnosis of new onset type 1 diabetes within 12 weeks of symptoms according to the American Diabetes Association (ADA) criteria.
3. History of at least one positive result on testing for any of the following antibodies: Islet-cell autoantibodies 512 (ICA512)/islet antigen-2 (IA-2), Glutamic Acid Decarboxylase (GAD) autoantibodies, Insulin autoantibodies.
4. Body weight > 30 kg.
5. Signs or symptoms of diabetes within 12 weeks of the first study visit.
6. Requires insulin > 0.2 units/kg body weight/day for T1DM
7. Fasting C-peptide greater than 0.3 ng/mL = 0.1 nmol/L = 100 pmol/L = 0.1 pmol/mL and Glucagon Stimulated C-peptide greater than 0.6 ng/mL = 0.2 nmol/L = 200 pmol/L = 0.2 pmol/mL.
8. Female of child bearing potential must have a negative pregnancy test and practice acceptable contraception [e.g., oral, intramuscular, or implanted hormonal contraception, sexual partner with nonreversed vasectomy (with azoospermia in 2 tests), 2 barrier methods (e.g., condom, diaphragm, or spermicide), or intrauterine device] or surgically sterile (tubal ligation or hysterectomy at least 6 months prior to first clinic visit)]. Female of childbearing potential must undergo pregnancy testing within 24 hours prior to administration of the first dose of study drug.
9. Able to swallow capsules.
10. Able to read, understand, and provide signed informed consent for the study (participants under the age of 18, shall provide an assent for the study as per country requirements).

Exclusion Criteria

Participants must not meet any of the following exclusion criteria to be eligible for the study:

1. Any medical condition that, in the opinion of the investigator, would interfere with safe completion of the trial or impact participant safety or evaluability of drug effect.
2. Prior administration of immunosuppressants at any time in the past, including in a clinical trial for type 1 diabetes.
3. Participation in any type of therapeutic drug or vaccine clinical trial within the last 12 weeks prior to the first clinic visit.
4. Taking any prescription medications, vitamins or herbal supplements that are contraindicated with cyclosporine within the last 14 days prior to first clinic visit.
5. Pregnant or lactating female.
6. Current therapy with GLP-1 receptor agonists (e.g., exenatide or pramlintide), or any other agents that might stimulate pancreatic beta cell regeneration or insulin secretion.
7. Current treatment with oral antidiabetic agents.
8. Evidence of active or latent tuberculosis.
9. Vaccination with a live virus or organism within the last 8 weeks prior to the first clinic visit.
10. Influenza vaccination with a killed virus, including booster vaccinations, within the last 4 weeks prior to the first clinic visit.
11. Vaccination with other antigens or killed organisms within the last 8 weeks prior to the first clinic visit.
12. Any infectious mononucleosis-like illness within the last 6 months prior to the first clinic visit.
13. History of or known active infection with HIV, HCV, or HBV.
14. Systolic or diastolic blood pressure >150 mmHg and > 90 mmHg, respectively, at the first clinic visit.
15. 95% percentile for weight at the first clinic visit.
16. An aspartate transaminase (AST), alanine transaminase (ALT), or total bilirubin level >2 times the upper limit of normal (ULN) at the first clinic visit.
17. A blood urea nitrogen (BUN) > 50 mg/dL (> 17.85 mmol/L) or a serum creatinine level > 1.3 mg/dL (> 115 µmol/L) at the first clinic visit.
18. A serum amylase level > 1.5 times the ULN or a serum lipase level > 2 times the ULN at the first clinic visit.
19. A history of substance abuse or dependence within the last 12 months prior to the first clinic visit as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM V) criteria.

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Insulin Independence and Hemoglobin A1c (A1C) < 6.5% | 24 weeks

SECONDARY OUTCOMES:
Safety and tolerability | 24 weeks
Pancreatic beta cell function measured by glucagon stimulated C-peptide response | 24 weeks
Proportion of participants achieving insulin independence | 24 weeks
Blood glucose control measured by A1C | 24 weeks
Average daily insulin requirement per week | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Professor Paolo Pozzilli, MD, Principal Investigator — Head, Endocrinology and Diabetes Unit, Campus Bio-Medico University of Rome

REFERENCES:
- [Background] Assan R, Blanchet F, Feutren G, Timsit J, Larger E, Boitard C, Amiel C, Bach JF. Normal renal function 8 to 13 years after cyclosporin A therapy in 285 diabetic patients. Diabetes Metab Res Rev. 2002 Nov-Dec;18(6):464-72. doi: 10.1002/dmrr.325. PMID 12469360
- [Background] Bougneres PF, Carel JC, Castano L, Boitard C, Gardin JP, Landais P, Hors J, Mihatsch MJ, Paillard M, Chaussain JL, et al. Factors associated with early remission of type I diabetes in children treated with cyclosporine. N Engl J Med. 1988 Mar 17;318(11):663-70. doi: 10.1056/NEJM198803173181103. PMID 3125434
- [Background] Eisenbarth GS Immunotherapy of diabetes and selected autoimmune diseases, CRC Press, Inc. 1989:61-72.
- [Background] Feutren G, Papoz L, Assan R, Vialettes B, Karsenty G, Vexiau P, Du Rostu H, Rodier M, Sirmai J, Lallemand A, et al. Cyclosporin increases the rate and length of remissions in insulin-dependent diabetes of recent onset. Results of a multicentre double-blind trial. Lancet. 1986 Jul 19;2(8499):119-24. doi: 10.1016/s0140-6736(86)91943-4. PMID 2873396
- [Background] Griffin KJ, Thompson PA, Gottschalk M, Kyllo JH, Rabinovitch A. Combination therapy with sitagliptin and lansoprazole in patients with recent-onset type 1 diabetes (REPAIR-T1D): 12-month results of a multicentre, randomised, placebo-controlled, phase 2 trial. Lancet Diabetes Endocrinol. 2014 Sep;2(9):710-8. doi: 10.1016/S2213-8587(14)70115-9. Epub 2014 Jul 2. PMID 24997559
- [Background] Jang JY, Kim SW, Han JK, Park SJ, Park YC, Joon Ahn Y, Park YH. Randomized prospective trial of the effect of induced hypergastrinemia on the prevention of pancreatic atrophy after pancreatoduodenectomy in humans. Ann Surg. 2003 Apr;237(4):522-9. doi: 10.1097/01.SLA.0000059985.56982.11. PMID 12677149
- [Background] Levetan C, Pozzilli P, Jovanovic L, Schatz D. Proposal for generating new beta cells in a muted immune environment for type 1 diabetes. Diabetes Metab Res Rev. 2013 Nov;29(8):604-6. doi: 10.1002/dmrr.2435. PMID 23853103
- [Background] Meier JJ, Ritzel RA, Maedler K, Gurlo T, Butler PC. Increased vulnerability of newly forming beta cells to cytokine-induced cell death. Diabetologia. 2006 Jan;49(1):83-9. doi: 10.1007/s00125-005-0069-3. Epub 2005 Dec 2. PMID 16323002
- [Background] Rigby MR. Non-immune-based treatment for type 1 diabetes: the way to go? Lancet Diabetes Endocrinol. 2014 Sep;2(9):681-2. doi: 10.1016/S2213-8587(14)70139-1. Epub 2014 Jul 2. No abstract available. PMID 24997558
- [Background] Singh PK, Hota D, Dutta P, Sachdeva N, Chakrabarti A, Srinivasan A, Singh I, Bhansali A. Pantoprazole improves glycemic control in type 2 diabetes: a randomized, double-blind, placebo-controlled trial. J Clin Endocrinol Metab. 2012 Nov;97(11):E2105-8. doi: 10.1210/jc.2012-1720. Epub 2012 Aug 17. PMID 22904177
- [Background] Skyler JS, Rabinovitch A. Cyclosporine in recent onset type I diabetes mellitus. Effects on islet beta cell function. Miami Cyclosporine Diabetes Study Group. J Diabetes Complications. 1992 Apr-Jun;6(2):77-88. doi: 10.1016/1056-8727(92)90016-e. PMID 1611143
- [Background] Sobel DO, Henzke A, Abbassi V. Cyclosporin and methotrexate therapy induces remission in type 1 diabetes mellitus. Acta Diabetol. 2010 Sep;47(3):243-50. doi: 10.1007/s00592-010-0188-2. Epub 2010 May 4. PMID 20440520
- [Background] Cyclosporin-induced remission of IDDM after early intervention. Association of 1 yr of cyclosporin treatment with enhanced insulin secretion. The Canadian-European Randomized Control Trial Group. Diabetes. 1988 Nov;37(11):1574-82. PMID 2903105
- See also: Related Info — http://www.nlm.nih.gov/medlineplus/diabetestype1.html